CLINICAL TRIAL: NCT01618890
Title: A Multi-center Randomized Controlled Study of Primary Prevention of Esophageal Variceal Bleeding in Cirrhotic Patients Treated With HVPG-guided Beta- Blocker Therapy or Standard Heart Rate-guided Beta-blocker Therapy
Brief Title: Hepatic Venous Pressure Gradient-guided Versus Standard Beta-blocker Therapy in Primary Prevention of Variceal Bleeding
Acronym: Porthos
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Free University Medical Center (Other); Haga Hospital (Other); Universitaire Ziekenhuizen KU Leuven (Other); Ziekenhuis Netwerk Antwerpen (ZNA) (Other)
Responsible Party: Principal Investigator, Dr. M.J.Coenraad, Dr., Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUMC-40226
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Acute Bleeding Esophageal Varices; Liver Cirrhosis
Keywords: Prevention; Esophageal variceal bleeding; Hepatic Venous Pressure Gradient; Betablocker therapy
MeSH Terms: conditions — Liver Cirrhosis | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HVPG-propranolol arm (Experimental): A baseline hepatic venous pressure gradient measurement (HVPG measurement) is performed in day-care setting. After this procedure propranolol is started at 20 mg BID. with dose escalation as described in the propranolol arm.
  A second HVPG measurement is performed at 4 weeks after adequate propranolol therapy. In patients who reach target HVPG reduction (responders), propranolol is continued at the same dose without routine control endoscopy. In patients who do not reach target HVPG reduction (nonresponders), endoscopic band ligation is performed in day-care setting with intervals of 2-4 weeks until complete obliteration of varices. Follow-up endoscopy with 6 months interval is performed to detect and treat recurrent large varices.
  Interventions: Procedure: Hepatic venous pressure gradient measurement
- Propranolol arm (No Intervention): Propranolol start 20 mg BID. orally with dose escalation based on heart frequency (HF) with 3-days interval to the maximum tolerated dose. No routine control endoscopy is required.

INTERVENTIONS:
Procedure: Hepatic venous pressure gradient measurement — Perform baseline HVPG measurement, then start propranolol 20 mg orally twice daily (BID), increase the dose stepwise to maximum tolerated dose. After 4 weeks a second HVPG is performed.
  In hemodynamic nonresponders from the study arm, repeated endoscopic band ligation is performed in daycare setting with intervals of 2-4 weeks.
  In hemodynamic responders (HVPG second measurement< 12 mmHg or >20% reduction in HVPG compared to baseline) beta-blockers are continued until end of follow-up.
  Other Names: Hepatic venous pressure measurement; Endoscopic variceal band ligation; Propranolol
  Arms: HVPG-propranolol arm

SUMMARY:
Study hypothesis:

Hepatic venous pressure gradient (HVPG)-directed primary prophylaxis with nonselective beta-blocker therapy (NSBB) leads to a reduction in first variceal bleeding episodes and is cost-effective in the long term.

Study design:

A multi-center randomized controlled study comparing nonselective beta-blocker therapy guided by the hemodynamic response as determined by the difference in HVPG before and after starting oral NSBB therapy, to standard heart rate-guided NSBB therapy in patients with esophageal varices due to liver cirrhosis without a history of esophageal variceal hemorrhage.

Primary study parameters/outcome of the study:

First variceal bleeding episodes occurring within the first two years.

Secondary study parameters/outcome of the study:

* Mortality
* Occurrence of other cirrhosis-related complications
* Occurrence of hepatocellular carcinoma
* Costs of treatments
* Adverse effects

DETAILED DESCRIPTION:
Background of the study:

About 50% of cirrhotic patients who use nonselective beta-blockers (NSBB) for primary prevention of variceal bleeding do not reach target hemodynamic response, defined as HVPG < 12 mmHg or a > 20% decrease in HVPG from baseline. These so-called hemodynamic nonresponding patients have significantly higher rate of first esophageal variceal hemorrhage as compared to patients who do respond to NSBB.

International institutions that publish guidelines differ in their recommendations concerning HVPG monitoring. As a result, practice currently varies widely.

The investigators hypothesize that HVPG-directed primary prophylaxis leads to a reduction in first variceal bleeding episodes and is cost-effective in the long term.

Objective of the study:

To determine cost-effectiveness of hepatic venous pressure gradient (HVPG)-guided nonselective beta-blocker therapy as compared to standard heart rate-guided beta-blocker therapy in the primary prevention of esophageal variceal bleeding in cirrhotic patients.

Study design:

A multi-center randomized controlled study comparing nonselective beta-blocker therapy guided by the hemodynamic response as determined by the difference in HVPG before and after starting oral nonselective beta-blockers, to standard heart rate-guided nonselective beta-blocker therapy in patients with esophageal varices due to liver cirrhosis.

Study population:

Patients with liver cirrhosis and large (>5 mm) esophageal varices without a history of esophageal variceal hemorrhage.

Intervention:

-In HVPG-group: Perform baseline HVPG measurement, then start propranolol 20 mg orally twice daily (BID), increase the dose stepwise with 3 days interval to decrease the heart rate to maximum tolerated dose. After 4 weeks a second HVPG is performed.

In hemodynamic responders (who reach target decrease in HVPG) NSBB are continued until end of follow-up.

In hemodynamic nonresponders (who do not reach target decrease in HVPG), NSBB are continued and repeated endoscopic band ligation is performed with 2-4 weeks interval until complete obliteration of large varices.

-In control group: Start propranolol 20 mg BID, increase the dose stepwise with 3 days interval to maximum heart rate-guided tolerated dose.

Primary study parameters/outcome of the study:

First variceal bleeding episodes occurring within the first two years.

Secondary study parameters/outcome of the study:

Mortality Occurrence of other cirrhosis-related complications Occurrence of hepatocellular carcinoma Costs of treatments Adverse effects

ELIGIBILITY:
Inclusion Criteria:

Patients with liver cirrhosis Large (≥5 mm) esophageal varices

Exclusion Criteria:

* History of esophageal variceal hemorrhage
* Pregnancy
* Contraindications to beta-blocker therapy
* Esophageal varices in the absence of liver cirrhosis
* Intermediate, advanced or terminal stage hepatocellular carcinoma (BCLC stage B, C or D)
* Refractory ascites
* Hepatorenal syndrome
* Prior treatment or prophylaxis for esophageal varices or varices bleeding (propranolol use, TIPS, endoscopic banding ligation, endoscopic sclerotherapy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2012-09 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
First variceal bleeding episodes | two years of follow-up
  First variceal bleeding episodes

SECONDARY OUTCOMES:
Mortality | two years
  Mortality
Occurrence of other cirrhosis-related complications | two years
  ascites spontaneous bacterial peritonitis hepatic encephalopathy hepatorenal syndrome hepatocellular carcinoma
Costs of treatments | two years
  Costs of treatments
Adverse effects | two years
  Adverse effects associated with NSBB therapy, endoscopic band ligation, hepatic venous pressure gradient

CONTACTS AND LOCATIONS:
Overall Officials: Minneke Coenraad, Dr., Principal Investigator — Leiden University Medical Centre
Locations (6):
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Universitaire Ziekenhuizen Leuven, Leuven
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam
  - Free University Medical Centre, Amsterdam
  - Leiden University Medical Centre, Leiden
  - Haga Hospital, The Hague